CLINICAL TRIAL: NCT06962449
Title: Analysis of Treatment Patterns and Clinical Outcomes After First-Line Treatment With Tislelizumab in Advanced NSCLC: A Real-World Observational Study
Brief Title: Real-World Assessment of Therapeutic Strategies and Survival Outcomes Following First-Line Tislelizumab Therapy in Advanced Non-Small Cell Lung Cancer
Acronym: REALM-Post
Status: Enrolling by invitation | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Tianqing Chu, Professor, Shanghai Chest Hospital
Other Study IDs: IS24123
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Non-Small-Cell Lung Cancer; Non-Small-Cell Lung Cancer Stage IV
Keywords: advanced non-small-cell Lung cancer; real-world study; Tislelizumab; progression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is an observational study evaluating the treatment patterns and clinical outcomes after progression on first-line Tislelizumab treatment in advanced NSCLC. Based on the inclusion and exclusion criteria, patients with advanced NSCLC who received first-line Tislelizumab treatment and progressed will be retrospectively screened and collected from January 1, 2020, to the study initiation date, and followed up for observation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable locally advanced or metastatic NSCLC based on the 8th edition of the AJCC staging system.
* Previously received first-line treatment with Tislelizumab for advanced NSCLC.
* Medical records of disease progression after first-line treatment.

Exclusion Criteria:

* Patients with incomplete key baseline and treatment information，including clinical stage, pathological type, treatment regimen, tumor assessment record after treatment ect.
* Patients included in anti-tumor drug intervention or unblinded clinical trials, in which the treatment being administered is unknown.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced NSCLC who progressed after first-line treatment with Tislelizumab
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
real-world progression-free survival | the time from the start of treatment to the first recorded progression event in the medical information system or death from any cause, whichever occurs first, excluding events within 14 days after the start of treament.
  rwPFS is defined as the time from the start of treatment to the first recorded progression event (imaging report or clinician judgment) in the medical information system or death from any cause, whichever occurs first, excluding events within 14 days after the start of treatment.
overall survival (OS) | From date of diagnosis until the date of death from any cause, whichever came first, assessed up to 60 months
  from diagnosis to death

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China